CLINICAL TRIAL: NCT01987466
Title: Plasma Neutrophil Gelatinase-associated Lipocalin (NGAL) as Early Biomarker for Renal Dysfunction and Good Neurologic Outcome in Out of Hospital Cardiac Arrest Patients
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Yonsei University (Other)
Responsible Party: Sponsor
Other Study IDs: 4-2013-0575
Record Dates: First submitted 2013-11-12; First posted 2013-11-19 (Estimated); Last update posted 2013-11-19 (Estimated); Status verified 2013-11

CONDITIONS: Post Cardiac Arrest Patient Who Was Treated by Hypothermia Protocol
Keywords: Neutrophil Gelatinase-associated Lipocalin(NGAL); Acute renal failure; Cardiac arrest; Hypothermia
MeSH Terms: conditions — Acute Kidney Injury; Heart Arrest; Hypothermia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Post cardiac arrest patient
  Interventions: Biological: Serum NGAL level

INTERVENTIONS:
Biological: Serum NGAL level — Investigators will check the plasma NGAL level after 4 hour from resuscitation. The plasma NGAL level is measured in ng/mg

SUMMARY:
Postresuscitation disease is a constellation of disorders related to whole-body ischemia and reperfusion syndrome. It includes hypoxic damage in brain, liver, kidney, heart and other organ. In previous study more than one-third of patients resuscitation from out of hospital cardiac arrest developed renal dysfunction. In acute kidney injury, NGAL is an earlier marker compared with serum creatinine.

Cardiac arrest and severe asphyxia result in global brain ischemia. In previous study serum NGAL correlated with hypoxic ischemic encephalopathy in asphyxiated neonate.

This study was designed to assess serum NGAL level in postresuscitative patients to evaluate its relation to hypoxic brain injury severity, and its clinical utility for early detection of acute kidney injury in these patients.

ELIGIBILITY:
Inclusion Criteria:

* 19 years and older
* Successful resuscitation from out of hospital cardiac arrest and spontaneous circulation time is longer than 20 min.
* GCS < 8

Exclusion Criteria:

* Pre-existing coma before cardiac arrest
* Mental change with other cause except cardiac arrest.(Ex. traumatic brain injury, cerebro-vascular accident.)
* Unstable vital sign (Systolic blood pressure is lower than 60mmHg)
* History of terminal illness.
* Coagulation deficiency.
* Pregnancy state or younger than 18 year
* Pre-existing end-stage renal disease or dependence on renal replacement therapy
* Transfer to other hospital and cannot know prognosis
* Withdrawal of care due to family wishes
* The patient arrives our hospital after 4 hours or longer from resuscitation.
* The patient refuses to sign the consent

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients over 19 years of age admitted to our hospital after succesful resuscitation from out of hospital cardiac arrest. Mental state of the patient is less than 8 in GCS scale and the patient should be undergoing therapeutic hypothermia.Exclusion criteria is age younger than 19 years, terminal illness or do-not resuscitation status, pre-existing coma, abnormal mental status with defined intracranial lesion (ex. cerebral hemorrhage, cerebral infarction, etc), unstable vital sign and previous end-stage renal disease.
Sampling Method: Non-Probability Sample
Enrollment: 73 (Estimated)
Dates: Start 2013-10; Primary Completion 2015-10 (Estimated); Study Completion 2015-10 (Estimated)

PRIMARY OUTCOMES:
Predictive value of plasma NGAL for acute kidney injury and cerebral dysfunction following out of hospital cardiac arrest. | Every 4 hour until 72 hour after resuscitation
  All patients in this study will be treated by induced hypothermia protocol in our hospital. Plasma NGAL level will check after 4hour from resuscitation. Renal dysfunction is defined using the RIFLE criteria. Patient base line creatinine is defined the first laboratory values obtained in the emergency department. The maximum difference between the peak creatinine level during the first 72hour of hospitalization and the base line creatinine level was determined for every patients.
  Cerebral dysfunction is defined using CPC scale. Neurologic exam will be performed on arrival, 24, 48,72 hours after resuscitation and discharge day. Good neurologic outcome is defined as CPC of 1 or 2. The diagnostic accuracy of NGAL in predicting acute kidney injury and neurologic outcome will be evaluated.

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Emergency Medicine, Severance Hospital, Yonsei University Health System, Seoul, South Korea

REFERENCES:
- [Derived] Lee JH, Park I, You JS, Kim MJ, Lee HS, Park YS, Park HC, Chung SP. Predictive performance of plasma neutrophil gelatinase-associated lipocalin for neurologic outcomes in out-of-hospital cardiac arrest patients treated with targeted temperature management: A prospective observational study. Medicine (Baltimore). 2019 Aug;98(34):e16930. doi: 10.1097/MD.0000000000016930. PMID 31441881